CLINICAL TRIAL: NCT03047668
Title: POLY-unsaturated Fatty Acids in the Preservation of Dietary Effects on Hepatosteatosis and Energy Metabolism in Type 2 Diabetes
Acronym: POLYPHEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Institute of Human Nutrition (Other)
Collaborators: German Center for Diabetes Research (Other); California Walnut Commission (Other); Institute for Cereal Processing GmbH/Institut für Getreideverarbeitung (IGV) (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas F. H. Pfeiffer, PI, German Institute of Human Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POLYPHEM
Record Dates: First submitted 2016-11-21; First posted 2017-02-09 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes; NAFLD; Obesity; Dyslipidemia; Hypertension; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease; Obesity; Dyslipidemias; Hypertension; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- low-carb with PUFA (Active Comparator): 49 weeks of hypo- to isocaloric low-carb diet (< 40 EI% carbs), amplified with walnuts and walnut-sunflower muffins
  Interventions: Dietary Supplement: diet with/without supplementation
- low-carb without PUFA (Active Comparator): 49 weeks of hypo- to isocaloric low-carb diet (< 40 EI% carbs), without walnuts / walnut-sunflower muffins
  Interventions: Dietary Supplement: diet with/without supplementation
- low-fat with PUFA (Active Comparator): 49 weeks of hypo- to isocaloric low-fat diet (< 30 EI% fat), amplified with walnuts and walnut-sunflower muffins
  Interventions: Dietary Supplement: diet with/without supplementation
- low-fat without PUFA (Active Comparator): 49 weeks of hypo- to isocaloric low-fat diet (< 30 EI% fat), without walnuts / walnut-sunflower muffins
  Interventions: Dietary Supplement: diet with/without supplementation

INTERVENTIONS:
Dietary Supplement: diet with/without supplementation — diet with/without supplementation with PUFAs

SUMMARY:
Basic treatment of type 2 diabetes should focus on diet, physical activity and lifestyle. Nevertheless, in early and late stage of T2DM, lifestyle intervention is mostly substituted by pharmacological intervention, although lifestyle modification and dietary treatment would be favourable.

The researchers therefore investigate dietary strategies such as low-carb and very-low calory diets regarding their potential to improve metabolism and body weight in (mostly) long-term T2DM patients. This core comparison is dealt with in the DiNA-D study (published elsewhere).

POLYPHEM targets specific dietary approach to preserve the achieved metabolic improvements from DiNA-D phase 1. Nutritional factors will be PUFAs and BCAAs.

DETAILED DESCRIPTION:
Basic treatment of type 2 diabetes should focus on diet, physical activity and lifestyle. Nevertheless, in early and late stage of T2DM, lifestyle intervention is mostly substituted by pharmacological intervention, although lifestyle modification and dietary treatment would be favourable.

The researchers therefore investigate dietary strategies such as low-carb and very-low calory diets regarding their potential to improve metabolism and body weight in (mostly) long-term T2DM patients. This core comparison is dealt with in the DiNA-D study (published elsewhere).

POLYPHEM targets specific dietary approach to preserve the achieved metabolic improvements from DiNA-D phase 1. Nutritional factors for the maintenance period within DiNA-D (11 months) will be PUFAs and BCAAs, provided by walnuts and custom-made muffins containing walnuts, sunflower oil and isomaltulose.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects
* 18-79 years old
* type 2 diabetes

Exclusion Criteria:

* renal insufficiency
* anaemia
* immunosuppression
* previous symptomatic cancer diagnosis
* acute cardiovascular disease (stroke, coronary syndrome)
* pregnancy and lactation
* severe psychiatric disorders
* corticoid or other immunosuppressive therapy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-05; Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
change in insulin secretion (glucagon stimulation test) | 49 weeks
  change in insulin secretion (glucagon stimulation test)
change in hepatic fat content (MR-S) | 49 weeks
  change in hepatic fat content (MR-S)
change in insulin secretion in the mixed-meal tolerance test (MMTT) - combined parameter | 49 weeks
  change in insulin secretion in the mixed-meal tolerance test (MMTT) - combined parameter
change in insulin sensitivity in the mixed-meal tolerance test (MMTT) - combined parameter | 49 weeks
  change in insulin sensitivity in the mixed-meal tolerance test (MMTT) - combined parameter
change in blood glucose profile in the mixed-meal tolerance test (MMTT) - combined parameter | 49 weeks
  change in blood glucose profile in the mixed-meal tolerance test (MMTT) - combined parameter

SECONDARY OUTCOMES:
inflammatory reaction in subcutaneous adipose tissue (SCAT analysis on protein and RNA level - IL-1; IL1beta, IL-6) | 49 weeks
  inflammatory reaction in subcutaneous adipose tissue (SCAT analysis on protein and RNA level - IL-1; IL1beta, IL-6)
change in parameters of peripheral neuropathy - vibration threshold | 49 weeks
  change in parameters of peripheral neuropathy - vibration threshold
change in parameters of peripheral neuropathy - thermal sensitivity | 49 weeks
  change in parameters of peripheral neuropathy - thermal sensitivity
change in parameters of peripheral neuropathy - pain thresholds | 49 weeks
  change in parameters of peripheral neuropathy - pain thresholds
change in parameters of autonomic neuropathy - measures of cardio-autonomic neuropathy (MSDD) | 49 weeks
  change in parameters of autonomic neuropathy - measures of cardio-autonomic neuropathy (MSDD)
change in parameters of autonomic neuropathy - measures of cardio-autonomic neuropathy (SANN) | 49 weeks
  change in parameters of autonomic neuropathy - measures of cardio-autonomic neuropathy (SANN)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas FH Pfeiffer, Prof. Dr. med., Principal Investigator — DIfE
Locations (1):
- DIfE (German Institute for Human Nutrition), Berlin, Germany